CLINICAL TRIAL: NCT01620359
Title: Study of ExAblate Focused Ultrasound Ablation of Breast Cancer Under MR Guidance (MRgFUS) and MRI Evaluation of Ablation
Brief Title: Study of ExAblate Focused Ultrasound Ablation of Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: InSightec (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BC006
Record Dates: First submitted 2012-06-13; First posted 2012-06-15 (Estimated); Last update posted 2016-08-31 (Estimated); Status verified 2016-08

CONDITIONS: Breast Cancer
Keywords: Breast cancer; Breast tumor; stage 1 disease; T1 M0 N0
MeSH Terms: conditions — Breast Neoplasms; Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ExAblate (Experimental)
  Interventions: Device: ExAblate MRgFUS

INTERVENTIONS:
Device: ExAblate MRgFUS — 100% ablation of an up-to-2-cm breast cancer visible on an contrast-enhanced MRI with 5-10 mm margins around the primary tumor

SUMMARY:
The goal of this prospective, non-randomized, single-arm, multi site, international study is to develop data to evaluate the safety and effectiveness of the ExAblate MRgFUS system in the ablation of breast cancer and of MRI.

The goal of MRgFUS ablation of breast cancer is to plan and ablate the entire tumor volume in a treatable and device accessible location.

DETAILED DESCRIPTION:
In this international, non-randomized, single-arm study, a total of 200 patients with a positive diagnosis of invasive breast cancer with a scheduled surgical resection will be enrolled into the trial. Eligible participants will be evaluated and treated with ExAblate breast ablation prior to their planned definitive surgical treatment. After the 10 to 21 days post ExAblate therapy, study participants will have another contrast-enhanced MR imaging examination. Their planned tumor excision will then be completed no later than 14 days from the contrast-enhanced, post ExAblate procedure MR imaging examination. Additionally, the end points of the study will be compared against the CORE Pathology Lab results.

ELIGIBILITY:
Inclusion Criteria:

1. Women age 18 years with invasive breast cancer
2. Patient with contrast-enhanced MR imaging confirming a single focal breast lesion less than 2 cm in diameter
3. Lesion clearly seen on contrast-enhanced MR and in a treatable location
4. Patient who is willing to undergo and be scheduled for sentinel lymph node biopsy
5. Patient scheduled and consented to surgical (lumpectomy or mastectomy) resection of the breast cancer
6. Patient with clinical Stage I disease: T1 M0 N0
7. Patient who signs an informed consent form for screening, SLNB, ablation, and follow-up visits.

Exclusion Criteria:

1. Invasive lobular carcinoma;
2. DCIS without invasive components on core biopsy;
3. Tamoxifen, Aromatase Inhibitors, and Neoadjuvant chemotherapy within 30 days prior to ExAblate.
4. Prior XRT or ablative therapy to the target breast;
5. Patients currently receiving anticoagulation therapy within the previous 14 days;
6. Lesions difficult to target (<1 cm from skin, nipple or the rib cage), as visualized on pre-therapy MRI;
7. Microcalcifications as the only sign of breast cancer on imaging studies;
8. Extensive intraductal components (EIC) on core biopsy.
9. Patients with breast implants;
10. Patients with prior surgical clips or other markers at the site of the breast tumor;
11. Patients with severe cerebrovascular disease (multiple CVA or CVA within 6 months);
12. hemolytic anemia (hematocrit < 30);
13. Pregnant or lactating, post-partum women;
14. Patient overall health status of ASA >2
15. Patient with active and ongoing infection at any body site;
16. Poor blood glucose control.
17. Severe hypertension
18. Patients with unstable cardiac status
19. Contraindication to MR or ExAblate ablation therapy
20. Patient with history of deep vein thrombosis
21. With history of pulmonary embolism;
22. Patient with sleep apnea;
23. Patient with airway problems;
24. Patient with severe claustrophobia;
25. Patient with non-MRI compatible implanted metal devices;
26. Patient with difficulty lying prone and still for up to 3 hours (180 minutes) in the MR unit;
27. Patient who cannot fit comfortably in the magnet or patients >250 lbs;
28. Patient with prior reaction to contrast agent;
29. Patient with history of grand mal seizures;
30. Patient with severely impaired renal function with estimated glomerular filtration rate <30 mL/min/1.73m2 and/or who is on dialysis;

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2011-06; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Adverse Events | 5 weeks post treatment
  To evaluate the incidence and severity of the ExAblate MRgFUS device-related complications to establish the safety profile of the ExAblate ablation of breast cancer visible on contrast-enhanced MRI with 5-10 mm margins around the primary tumor
Histopathological analyses | 5 weeks post treatment
  To estimate the effectiveness of ExAblate MRgFUS to ablate 100% of an up-to-2-cm breast cancer visible on an contrast-enhanced MRI with 5-10 mm margins around the primary tumor.

SECONDARY OUTCOMES:
MR imaging | 5 weeks post treatment
  To estimate the sensitivity of post-ablation MRI in identifying residual disease following ablation.

CONTACTS AND LOCATIONS:
Overall Officials: Hans Kolberg, MD, Principal Investigator — FUS BOTTROP
Locations (1):
- Marienhospital, Bottrop, Germany

REFERENCES:
- See also: Sponsor's website — http://WWW.INSIGHTEC.COM